CLINICAL TRIAL: NCT01451034
Title: Clinical Outcomes of Endoscopic Resection for Treating Extremely Well Differentiated Intestinal-type Adenocarcinoma (WHYX Lesion)
Brief Title: Clinical Outcomes of Endoscopic Resection for Treating WHYX Lesion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-08-022
Record Dates: First submitted 2011-09-28; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: WHYX Lesion; Extremely Well Differentiated Intestinal-type Adenocarcinoma
Keywords: WHYX lesion; endoscopic resection; complete resection; complete resection rate; endoscopic feature; Average size discrepancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WHYX cancer group (Active Comparator): WHYX cancer diagnosed by pathologic report
  Interventions: Procedure: WHYX cancer group
- non-WHYX cancer group (Placebo Comparator): all cancer except WHYX cancer diagnosed by pathologic report
  Interventions: Procedure: WHYX cancer group

INTERVENTIONS:
Procedure: WHYX cancer group — WHYX cancer diagnosed by pathologic report

SUMMARY:
Endoscopically, WHYX cancers demonstrated a vague extent of tumor spread due to pale color changes in both the background atrophic and metaplastic gastric mucosa. However, the clinical outcomes of WHYX cancers after endoscopic resection are unknown. The aim of this study was to evaluate clinical outcomes of WHYX cancers after endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

* From January 2009 to December 2010 enrolled 872 patients with EGC

Exclusion Criteria:

* EGC with regional lymph node metastasis in radiologic finding endoscopically suspicious submucosal invasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
complete resection rate | 6 months after endoscopical resection
  Complete resection was defined to have all of the following features: 1. grossly en bloc resection, 2. Tumor-free lateral and vertical resection margins, 3. No lymphovascular invasion, and 5. A depth of submucosal tumor invasion of less than 500 micrometers.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea